CLINICAL TRIAL: NCT06792149
Title: Research on the Value of Predicting Drug Efficacy Based on 3D Bioprinting for Constructing In Vitro Gastric Cancer Models
Brief Title: Prediction of Drug Response in Gastric Cancer Based on 3D Bioprinting
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GC-3D-Bioprinting
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-06

CONDITIONS: STOMACH NEOPLASM
MeSH Terms: conditions — Stomach Neoplasms | interventions — Chemotherapy, Adjuvant; Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — resected tumor tissue from surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group A: gastric cancer patients at resectable stage II/III who will receive adjuvant chemotherapy after surgery
  Interventions: Procedure: surgical resection; Other: Adjuvant chemotherapy
- Group B: gastric cancer patients at locally advanced stage who will receive neoadjuvant chemotherapy before surgery and adjuvant chemotherapy after surgery
  Interventions: Procedure: surgical resection; Other: Adjuvant chemotherapy; Other: neoadjuvant therapy
- Group C: Gastric cancer patients who are not scheduled to undergo neoadjuvant chemotherapy prior to surgical intervention and who will not receive adjuvant chemotherapy during the postoperative follow-up period.
  Interventions: Procedure: surgical resection

INTERVENTIONS:
Procedure: surgical resection — Surgical resection will be performed for locoregional lesions .
Other: Adjuvant chemotherapy — Regimens of adjuvant chemotherapy are directed by clinical guidance and experience.
  Groups: Group A; Group B
Other: neoadjuvant therapy — Regimens of neoadjuvant chemotherapy are directed by clinicalguidance and experience
  Groups: Group B

SUMMARY:
The therapeutic regimens for adjuvant and neoadjuvant chemotherapy in gastric cancer (GC) predominantly hinge on clinical experience. Consequently, there is an imperative need for preclinical models to facilitate the guidance of individualized medicine. The investigators plan to establish three-dimensional (3D) bioprinted GC models derived from surgically resected tumor tissues of GC patients. These in vitro 3D models will be subjected to treatment with the identical chemotherapy drugs administered to the corresponding patients from whom the models are sourced. The sensitivity of the chemotherapy drugs will be assayed within the in vitro models, and the actual response to chemotherapy in patients will be meticulously evaluated. This observational study aims to substantiate the potential utility of 3D bioprinted tumor models in prognosticating the response to chemotherapy in GC.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* Patients previously diagnosed with gastric cancer or confirmed by pathology as having gastric cancer postoperatively.
* Patients who have undergone preoperative imaging examinations, including plain and contrast-enhanced CT scans of the chest, abdomen, and pelvis, as well as gastric MRI for tumor staging, and who are planned for preoperative (neo)adjuvant therapy after multidisciplinary team (MDT) discussion; patients with advanced gastric cancer who are confirmed by postoperative pathology to require (neo)adjuvant therapy.
* The patient or their family members are able to comprehend the research protocol and are willing to participate in this study, providing written informed consent.

Exclusion Criteria:

* History of other malignancies or serious medical conditions
* Inability to provide independent informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with a clinical and pathological diagnosis of gastric cancer are deemed eligible for this study. Clinical physicians will meticulously record the medical histories, restricting inclusion to patients aged 18 years and above. Exclusion criteria encompass individuals with concomitant malignancies or severe comorbidities. Patients incapable of providing autonomous informed consent are ineligible for participation. All participants will undergo adjuvant or neoadjuvant chemotherapy, followed by surgical resection, as part of the treatment protocol for localized gastric cancer.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of Drug Sensitivity in In Vitro Tumor Models with Clinical Response in Patients | From enrollment to end within 2 weeks
  1. Response of 3D tumor models to chemotherapy drugs identical to those administered to corresponding patients: Researchers will establish and culture 3D printed gastric cancer models and treat them with the same chemotherapy drugs used for the corresponding patients. Following treatment, the viability of the 3D tumor models will be observed, and the IC50 of each drug will be calculated. The correlation between the sensitivity of the 3D models and the patients' responses will be analyzed.
  2. Response of Gastric Cancer Patients to Neoadjuvant Chemotherapy: For patients who undergo neoadjuvant chemotherapy prior to surgery, the response to such treatment will be assessed based on clinical imaging results, the Mandard-TRG criteria, and the RECIST score.

SECONDARY OUTCOMES:
Response of Gastric Cancer Patients to Adjuvant Chemotherapy | Up to 2 years
  The response to adjuvant chemotherapy will be assessed based on disease-free survival (DFS) or Overall Survival (OS). Regular follow-ups will be conducted. DFS is defined as the interval between the date of surgery and the date of the last follow-up or the date of recurrence/progression.Overall survival (OS) is delineated as the temporal span from the date of surgery to the date of death or the date of the last follow-up, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) can be accessed with reasonable requests via e-mail. IPD will be shared after the study is completed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD data will available after the study is completed
Access Criteria: Data can be accessed via e-mail with reasonable requests.

REFERENCES:
- [Background] Yan HHN, Siu HC, Law S, Ho SL, Yue SSK, Tsui WY, Chan D, Chan AS, Ma S, Lam KO, Bartfeld S, Man AHY, Lee BCH, Chan ASY, Wong JWH, Cheng PSW, Chan AKW, Zhang J, Shi J, Fan X, Kwong DLW, Mak TW, Yuen ST, Clevers H, Leung SY. A Comprehensive Human Gastric Cancer Organoid Biobank Captures Tumor Subtype Heterogeneity and Enables Therapeutic Screening. Cell Stem Cell. 2018 Dec 6;23(6):882-897.e11. doi: 10.1016/j.stem.2018.09.016. Epub 2018 Oct 18. PMID 30344100
- [Background] Zhao Y, Li S, Zhu L, Huang M, Xie Y, Song X, Chen Z, Lau HC, Sung JJ, Xu L, Yu J, Li X. Personalized drug screening using patient-derived organoid and its clinical relevance in gastric cancer. Cell Rep Med. 2024 Jul 16;5(7):101627. doi: 10.1016/j.xcrm.2024.101627. Epub 2024 Jul 3. PMID 38964315